CLINICAL TRIAL: NCT00495365
Title: Evaluation of Dose Conversion From Variable Dosing Intervals of Darbepoetin Alfa to Variable Dosing Intervals of Epoetin Alfa in Patients With the Anemia of Chronic Kidney Disease
Brief Title: A Dose Conversion Study of Epoetin Alfa in Subjects With the Anemia of Chronic Kidney Disease.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was stopped due to slow enrollment
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005104
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Chronic Renal Insufficiency
Keywords: Anemia; low blood count; chronic kidney disease; chronic kidney failure; darbepoetin alfa; epoetin alfa; recombinant human erythropoietin
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study was to evaluate hemoglobin stability in subjects who had received darbepoetin alfa for a minimum of 3 months prior to study entry who were then converted to epoetin alfa at the same dosing frequency to maintain a hemoglobin level of 12 plus or minus 1 g/dL (range 11-13- g/dL).

DETAILED DESCRIPTION:
This was a prospective, multicenter study in subjects with chronic kidney disease. The study was designed to address hemoglobin stability after drug conversion to epoetin alfa in subjects previously receiving darbepoetin alfa therapy.

The study was to enroll approximately 180 subjects with chronic kidney disease. Eligible subjects were those with chronic kidney disease who were receiving darbepoetin alfa every two, three, or four weeks for a period of 3 months or more and who had a stable hemoglobin (Hb) level at study entry of 12 g/dL (plus or minus 1 g/dL (11-13 g/dL). Subjects receiving darbepoetin alfa every 2, 3 or 4 weeks were switched over to epoetin alfa which they received at the same dosing frequency ( every 2, 3 or 4 weeks) upon study entry and throughout the 24 week study period. Clinical safety was assessed for the occurrence and severity of adverse events. Blood tests (Complete Blood Count, platelets, reticulocyte count, iron, were assessed at pre-determined intervals throughout the study. Vital signs (e.g. Blood pressure) were checked at each visit. Subjects received epoetin alfa at the same dosing frequency that they had previously received darbepoetin alfa. Subjects received 20,000 Units (U) epoetin alfa subcutaneously (SC) every two weeks; 30,000 U epoetin alfa SC every 3 weeks; or 40,000 U epoetin alfa SC every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic kidney disease defined as serum creatinine of 1.5 to 6.0 mg/dL for women and 2.0 to 6.0 mg/dL for men
* glomerular filtration rate (GFR) within 15-60 mL/min
* Subjects on darbepoetin alfa for 3 months or more and with a stable entry hemoglobin level of 12 (plus or minus 1 g/dL
* range 11-13 g/dL)
* Subjects receiving darbepoetin alfa on an every two, three, or four week dosing schedule
* female subjects with a reproductive potential must have a negative ruine pregnancy test within 7days of the first dose of study drug.

Exclusion Criteria:

* No uncontrolled high blood pressure as assessed by the primary physician
* No known hypersensitivity to mammalian cell-derived products
* No known hypersensitivity to human albumin
* Not receiving dialysis or scheduled to receive dialysis during the course of the study
* No severe congestive heart failure (New York Heart Association Class IV)
* No known severe stable or unstable coronary artery disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-06; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
The primary objective was to evaluate the proportion of subjects who maintained hemoglobin levels within 10% of entry levels and/or a range of 11-13 g/dL for the 24-week duration of the study.

SECONDARY OUTCOMES:
The secondary objective was to evaluate safety in subjects with chronic kidney disease throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- See also: Evaluation of Dose Conversion from Variable Dosing Intervals of Darbepoetin Alfa to Variable Dosing Intervals of Epoetin Alfa (PROCRIT) in Patients with the Anemia of Chronic Kidney Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=927&filename=CR005104_CSR.pdf